CLINICAL TRIAL: NCT01264848
Title: Endovascular Correction of Chronic Cerebrospinal Venous Insufficiency (CCSVI) and Evaluation of Influence of These Treatments on the Symptoms of Multiple Sclerosis
Brief Title: Endovascular Treatment for Chronic Cerebrospinal Venous Insufficiency (CCSVI)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Euromedic Specialist Clinics, Poland (Other)
Responsible Party: Principal Investigator, Marian Simka, PhD, Euromedic Specialist Clinics, Poland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7/2010
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; venous insufficiency
MeSH Terms: conditions — Multiple Sclerosis; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon angioplasty and/or stenting (Experimental): Balloon angioplasty and/or stenting of stenosed internal jugular vein and/or azygous vein and/or brachiocephalic vein
  Interventions: Procedure: balloon angioplasty and/or stenting

INTERVENTIONS:
Procedure: balloon angioplasty and/or stenting — balloon angioplasty and/or stenting of internal jugular veins and/or azygous vein and/or brachiocephalic veins
Procedure: balloon angioplasty and/or stenting — balloon angioplasty and/or stenting of extracranial vein draining the central nervous system, on condition that such outflow pathology has been confirmed using catheter venography

SUMMARY:
The aim of this study is to assess the efficacy of endovascular treatment (balloon angioplasty and/or stenting) for the improvement of clinical symptoms in multiple sclerosis patients.

DETAILED DESCRIPTION:
The aim of this study is to assess the efficacy of endovascular treatment (balloon angioplasty and/or stenting) for the improvement of clinical symptoms in multiple sclerosis patients measured by Extended Disability Severity Score (EDSS), Multiple Sclerosis Impact Scale-29 (MSIS-29), Fatigue Severity Scale (FSS) and heat intolerance

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically defined multiple sclerosis

Exclusion Criteria:

* contraindication for endovascular procedure performed in local anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in clinical symptoms of multiple sclerosis measured by Extended Disability Severity Score (EDSS), Multiple Sclerosis Impact Scale-29 (MSIS-29), Fatigue Severity Scale (FSS) and heat intolerance | 6 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marian Simka, Principal Investigator — Euromedic Specialist Clinics , Katowice , Poland
Locations (1):
- Euromedic Specialist Clinics, Katowice, Poland